CLINICAL TRIAL: NCT00814151
Title: Primary Investigation Into the Performance of the MicroPhage S. Aureus / MSSA / MRSA Test Direct From Blood Culture.
Brief Title: MicroPhage S. Aureus / MSSA / MRSA Blood Culture Beta Trial
Status: Completed | Type: Observational
Sponsor: MicroPhage, Inc. (Industry)
Responsible Party: Scott Conlin, MicroPhage, Inc.
Other Study IDs: MP-2008B
Record Dates: First submitted 2008-12-22; First posted 2008-12-24 (Estimated); Last update posted 2008-12-24 (Estimated); Status verified 2008-12

CONDITIONS: Bacteremia; Staphylococcal Infection; Sepsis; Infection
Keywords: Blood culture; Staphylococcus aureus; Bacteremia; MRSA; MSSA; MicroPhage
MeSH Terms: conditions — Bacteremia; Staphylococcal Infections; Sepsis; Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Retention of discrepant blood culture specimens only.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MicroPhage: Blood Culture positive specimens available within 24 hours of alarm.
  Interventions: Other: MicroPhage S. aureus / MSSA / MRSA Blood Culture Test (prototype)
- Standard of Care: Blood Culture positive specimens.

INTERVENTIONS:
Other: MicroPhage S. aureus / MSSA / MRSA Blood Culture Test (prototype) — In vitro diagnostic: The MicroPhage "Intervention" was to perform the MicroPhage diagnostic test to detect S. aureus in the blood culture sample and determine MSSA or MRSA status at 4 and 5 hours of test incubation. The "Intervention" results were not made available to the patient or their physician.
  Groups: MicroPhage

SUMMARY:
In-vitro identification of S. aureus, methicillin-sensitive S. aureus (MSSA), and methicillin-resistant S. aureus (MRSA) from positive blood cultures by MicroPhage's bacteriophage-based diagnostic platform.

DETAILED DESCRIPTION:
This is a multi-center, preclinical study to investigate the effectiveness of the performance of MicroPhage S. aureus / MSSA/MRSA test direct for blood culture. There will be no patient consent, as this is a laboratory performance study on leftover specimens. The MicroPhage test will be compared to site standards (gold standard) and market-available tests with similar indications (comparators). MicroPhage will require data to be collected at 4 hours and 5 hours following the start of the MicroPhage test. The study will last 2-3 months, depending on the accrual rate of the institution.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Blood culture positive, of ANY of the following bottle types:
* BD Bactec Standard Aerobic and Anaerobic,
* BD Bactec Plus Aerobic and Anaerobic,
* bioMerieux BacT/Alert Standard Aerobic and Anaerobic,
* bioMerieux BacT/Alert FAN Aerobic and Anaerobic.

Exclusion Criteria:

* BD Bactec Lytic, Pediatric, or other bottle types not listed above.
* bioMerieux Pediatric FAN or other bottle types listed above.
* Trek bottles.
* Specimens from patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Blood culture positive specimens from three academic medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 712 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Determination of clinical performance of preliminary MicroPhage S. aureus/MSSA/MRSA test directly from clinical blood culture positives. | Within 48 hours

SECONDARY OUTCOMES:
Qualitative feedback on the preliminary MicroPhage test protocol.
Comparative results to market-available S. aureus / MRSA tests for Blood Culture. | Within 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: J D Smith, Ph.D., Principal Investigator — MicroPhage, Inc.
Locations (3):
- United States (3):
  - Evanston Northwestern Healthcare Research Institute, Evanston, Illinois
  - University of Maryland Baltimore, Baltimore, Maryland
  - Johns Hopkins Medical Institute, Baltimore, Maryland